CLINICAL TRIAL: NCT03220061
Title: Effectiveness of Music Therapy on Blood Pressure and Anxiety Among Patients Undergoing Haemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, ANU RANI PANCHAL, student, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200197
Record Dates: First submitted 2017-07-10; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: music therapy was soft and relaxing instrumental piano music which was given among haemodialysis patients for 30 minutes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): music therapy was used in the study for 30 minutes
  Interventions: Behavioral: music therapy
- control (No Intervention): usual care was given to participant in control group

INTERVENTIONS:
Behavioral: music therapy
  Arms: experimental

SUMMARY:
Effectiveness of music therapy on blood pressure and anxiety among patients undergoing haemodialysis

DETAILED DESCRIPTION:
Abstract Introduction:- dialysis is one of the technological innovation in medicine in which patients are being reported to face psychosocial and physiological problems such as anxiety, stress and hypertension etc. To relieve these problems, music therapy has been widely used as a non-pharmacological intervention with the aim to assess the effectiveness of music therapy on blood pressure and anxiety among haemodialysis patients.

Methods:- current study using true experimental pre-test post-test design was conducted among 60 haemodialysis patients which were randomly allocated to experimental (30) and control (30) group using simple random sampling. The data was collected through sample characteristics performa, blood pressure monitoring data sheet and beck anxiety inventory. Patients in experimental group were provided with 30 minutes of music therapy using slow and calm relaxing instrumental piano music whereas in control group only usual care was given.

ELIGIBILITY:
Inclusion Criteria:

* willing to participate in study
* alert, oriented and able to comprehend, speak and listen Hindi or English language.

Exclusion Criteria:

* altered sensorium
* hypotension
* unresponsiveness
* hearing disabilities

Ages: 17 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-12 (Actual)

PRIMARY OUTCOMES:
beck anxiety inventory | 10 minutes
  minimum score was 1 and maximum score was 63

CONTACTS AND LOCATIONS:
Overall Officials: anu R panchal, nursing, Principal Investigator — maharishi markandeshwar university
Locations (1):
- Maharishi Markandeshwar University, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
master data sheet
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: only publication
URL: http://anupanchal766@gmail.com